CLINICAL TRIAL: NCT03852186
Title: Towards Personalized Medicine for OCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Sara Kerstine Kaya Nielsen, Postdoctoral Researcher, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VD-2018-376
Record Dates: First submitted 2019-02-18; First posted 2019-02-25 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2019-02

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cognitive Behavioral Therapy; Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: Multicenter Non-inferiority Block Randomized Controlled Trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessor blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive behavioral therapy (Active Comparator): Manualized group-based cognitive behavioual therapy delivered by clinical psychologists and psychiatrists. The treatment consists of 14 sessions of each 2 hours.
  Interventions: Behavioral: Cognitive behavioral therapy
- Acceptance and commitment therapy (Experimental): Manualized group-based Acceptance and Commitment therapy delivered by clinical psychologists and psychiatrists. The treatment consists of 14 sessions of each 2 hours.
  Interventions: Behavioral: Acceptance and commitment therapy

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — Group based psychotherapy
  Arms: Cognitive behavioral therapy
Behavioral: Acceptance and commitment therapy — Group based psychotherapy
  Arms: Acceptance and commitment therapy

SUMMARY:
Obsessive compulsive disorder (OCD) is one of the most disabling anxiety disorders occurring in about 2 out of a 100 adults. Untreated, OCD is a chronic and deteriorating condition, negatively impacting multiple areas of life with high personal and socioeconomic costs. In Denmark, anxiety disorders are estimated to be the most expensive of all psychiatric disorders and the most common reason for forced retirement.

In many countries including DK, CBT is the recommended, first-line treatment for OCD. All individuals who seek treatment in the Danish Regions are offered CBT. However, reviews show that up to 50% of patients either do not respond to CBT or terminate treatment prematurely. Despite this large number of non-responders, no significant progress for OCD treatment has been made since initial efficacy trials. Alternatives to CBT are needed .

Acceptance and Commitment therapy (ACT) is an innovative psychotherapy that can potentially help individuals with OCD who do not benefit from CBT. ACT targets the habitual thinking and behaviors that mark OCD by aiming to increase value-based behavior. OCD often co-occurs with depression and other anxiety disorders making treatment more difficult. ACT is a transdiagnostic treatment targeting symptoms that are common to anxiety and mood disorders. Preliminary findings indicate that ACT may be an effective treatment for OCD. However, these findings constitute a low level of evidence. Before ACT can be declared as an effective treatment for OCD, it needs to be demonstrated in randomize controlled trials, in which ACT is compared to legitimate, active treatments, such as CBT. This project will test the effectiveness of group-based ACT by comparing it to the first-line treatment, group-CBT in 180 participants referred for treatment in a specialized outpatient clinic at the Mental Health Services, Capital Region of Denmark. Furthermore, moderators and predictors of treatment response will be investigated.

DETAILED DESCRIPTION:
Introduction Anxiety disorders are some of the most prevalent mental illnesses affecting 350.000-400.000 Danes every year. Obsessive compulsive disorder (OCD) is one of the most disabling anxiety disorders and is characterised by the presence of intrusive thoughts, urges, or images that cause anxiety, and, in turn, by repetitive behaviours that are often performed in an attempt to reduce the anxiety. OCD has a lifetime prevalence of 2-3 %. If left untreated, OCD is a chronic anxiety disorder resulting in deteriorating mental health with high personal costs and negative impacts on multiple areas of life. OCD is also associated with more functional impairment, more use of healthcare services and poorer quality of life than seen for any other patient group (including substance abuse and somatic illnesses). Additionally, OCD often precedes the onset of other common comorbid anxiety, mood, eating and substance abuse disorders and is strongly associated with suicide. The negative impact of OCD carries over into the families of patients and to society at large. In Denmark, anxiety disorders are estimated to be the most expensive of all disorders with annual costs estimated at 9.4 billion DKK, and they are the most common reason for forced retirement. The high personal and societal costs of OCD makes it a significant public health concern. Despite having been conceptualized as an illness with a poor prognosis, systematic reviews have consistently shown that cognitive behavioral therapy (CBT) including exposure and response prevention (ERP) is an effective treatment for OCD. This has made CBT the first choice for treating OCD in many mental health settings, as also recommended by the Danish Health Authorities. Nonetheless, a relatively large group of OCD patients does not benefit from CBT. Reviews of CBT-based treatment studies show that up to 50% of patients do not respond to CBT or terminate treatment prematurely. Despite the large number of non-responders, no significant progress for OCD treatment has been made since initial efficacy CBT trials in the 1970´ies. Thus, it is crucial to establish more effective psychotherapies (for the non-responders of CBT-based treatments) for OCD. Preliminary findings suggest that Acceptance and Commitment therapy (ACT) may be an effective treatment for OCD. ACT aims at increasing the participants valued actions in life (e.g. family life, work, sports), and the willingness to experience unpleasant emotions and thoughts. Both aspects are especially relevant for individuals with OCD, as a substantial amount of time is spent on OCD-behavior and avoiding the experience of distress and anxiety. To date, the support for ACT stems from smaller case studies and one controlled trial comparing ACT to Progressive Muscle Relaxation (PMR), including 79 individuals with OCD. The case studies showed that ACT was effective for OCD, and these positive results were also found in the controlled trial showing an effect size of 0.77 at post-treatment and of 1.10 at follow-up (3-months). Of the participants randomized to ACT, 46% showed significant symptom change compared to 13% of the participants who received PMR. Importantly, participants rated ACT as highly acceptable. However, serious limitations of the currently available evidence limit the conclusions that can be drawn on the effectiveness of ACT for OCD. First, the studies included relatively small samples. Second, PMR has not shown to be an effective treatment for OCD. Third, none of the previous studies have investigated the long-term effect of ACT on OCD. Thus, studies including a large sample and comparing the effect of ACT to the gold standard treatment, CBT, is warranted. Furthermore, studies should examine the long-term effect of ACT. In addition, previous studies have primarily been conducted in laboratory settings with maximal exclusion criteria which compromises the external validity. But OCD is commonly seen with comorbid depression and/or other anxiety diagnoses, so results based on highly selected patient samples treated in research clinics that specialize in OCD treatment are not generalizable to typical individuals with OCD or to clinics which treat most OCD patients. In sum, controlled trials comparing the effectiveness of ACT to CBT are warranted to confirm whether ACT is indeed the sought-after alternative to CBT.

What treatment works for whom? Another crucial step in order to improve the treatment for OCD is to consider individual patient characteristics in the composition of optimal treatment setups facilitating personalized treatment. This requires extensive knowledge of predictors and moderators of OCD treatment success. However, to date no reliable predictors or moderators have been identified. Previous predictor and moderator studies have suggested that attachment patterns and anxiety sensitivity may be related to treatment outcome for ACT and CBT. Accumulating studies also highlights the relevance of investigating biological markers in relation to OCD. However, very little is known about the role of biomarkers in OCD and in psychotherapy although studies are emerging.

Purpose This study aims to test the (long-term) effectiveness of ACT for OCD and to compare the effectiveness to CBT in a naturalistic clinical setting. Additionally, the aim is to identify reliable markers to guide efficient treatment choice by examining several theory-driven, putative predictors and moderators: 1) moderators which are theoretically connected to the two treatments (e.g. thought-action-fusion, anxiety sensitivity) 2) personality and interpersonal characteristics involved in the maintenance of OCD (e.g. emotion regulation, attachment style, personality traits) and 3) biomarkers known to be associated with comorbidity, chronicity and treatment refractivity. Finally, 4) the study will investigate the moderating effects of clinical and demographic characteristics (e.g. comorbid depression, gender, education, age). Main hypotheses 1: In the overall sample, both the ACT and CBT treatment will yield clinically significant results, indicated by a change in Yale-Brown Obsessive Compulsive Scale (Y-BOCS) scores from pre- to posttreatment, with ACT and CBT being equally effective. 2: The effect at 6- and 12-months follow-up will be equal for ACT and CBT, measured with Y-BOCS. 3: Participants with comorbid depression at baseline will benefit more from ACT than CBT. Method The study is a single blinded, pragmatic, non-inferiority, parallel, multi-center block randomized controlled trial of ACT vs CBT for OCD. In total, 180 patients are recruited from two regional MHS centers across Capital Region of Denmark and included in two intervention arms. The participants will be assessed with diagnostic interview and self-report measures at baseline, post-treatment, 6-months and 12-months follow-up. Randomization The randomization will be carried out based on an allocation list with permuted blocks using the Region´s secure system REDcap by a person not attached to the project.

Data analysis

Longitudinal data will be analyzed using Mixed Model Repeated Measures (MMRM) and Hierarchical Linear Modeling (HLM) and an intend-to-treat sample including all randomized participants. Detection of the moderating value of the proposed variables will be analyzed in the two domains, using the method proposed by Kraemer. The possible moderators will be examined for individual effect sizes and then entered into a forward-stepwise regression model predicting differential treatment response. K-fold cross validation will be used to identify the number of variables to be included in the final moderator model in order to identify moderators in rank-order. Timeplan The project is planned to start in January 2019 and will run over 4 years.

ELIGIBILITY:
Inclusion Criteria:

* have OCD as their primary diagnosis
* are between 18-65 years
* are free of alcohol and substance abuse
* are not receiving any other psychotherapy during the study
* are medication-free or stabilized on psychotropic medication
* speak and understand Danish
* provide written consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2019-03-02 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Yale Brown obsessive compulsive scale | 25 minutes
  Semi-structured interview, total score consists of all items of all items summed up, likert scale minimum 0- maximum 4, higher values predict worse OCD-symptoms
Quality of Life Inventory | 20 minutes
  Self-report measure, 16 items, minimum -3 - maximum 3. Higher scores indicate higher quality of life.
  measuring outcome in terms of an overall life satisfaction score, likert scale 0-6

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No